CLINICAL TRIAL: NCT00907621
Title: Effects of Acupuncture in the Treatment of Infant Colic: A Prospective Multi-center Single Blinded Randomized Controlled Study
Brief Title: Effects of Acupuncture in the Treatment of Infant Colic
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Oslo (Other)
Responsible Party: Principal Investigator, Arne Fetveit, Associate Professor, University of Oslo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: infant colic
Record Dates: First submitted 2009-05-21; First posted 2009-05-22 (Estimated); Results first posted 2015-03-17 (Estimated); Last update posted 2015-03-17 (Estimated); Status verified 2015-03

CONDITIONS: Infant Colic
Keywords: Infant Colic; Acupuncture; General Practice
MeSH Terms: conditions — Colic | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Acupuncture (Experimental): Acupuncture with Seirin 020x15 mm sterile acupuncture needle:
  Bilateral insertion of a Seirin 020x15mm sterile acupuncture needle to a depth of 12mm for 30 seconds during 3 consecutive working days at the WHO designated acupuncture point St36 on infants born after 36th week of gestation and weighing over 2500 grams at birth, and who qualify according to Wessels definition:
  Paroxystical, uncontrolled crying in an otherwise healthy child under 3 months of age, and with more than 3 hours of crying 3 days per week for 3 weeks.
  Interventions: Procedure: Acupuncture with Seirin 020x15 mm sterile acupuncture needle
- Control (No Intervention): Infants born after 36th week of gestation and weighing over 2500 grams at birth, and who qualify according to Wessels definition:
  Paroxystical, uncontrolled crying in an otherwise healthy child under 3 months of age, and with more than 3 hours of crying 3 days per week for 3 weeks.
  The Control group will have no intervention.

INTERVENTIONS:
Procedure: Acupuncture with Seirin 020x15 mm sterile acupuncture needle — Bilateral insertion of a Seirin 020x15mm sterile acupuncture needle to a depth of 12mm for 30 seconds during 3 consecutive working days at the WHO designated acupuncture point St36.
  Other Names: Seirin 020x15mm sterile acupuncture needle
  Arms: Acupuncture

SUMMARY:
Standardized acupuncture treatment for infant colic is a common treatment in general practice for doctors educated in medical acupuncture.

The investigators plan to study whether the perceived opinion on positive results can be verified in a multi-center clinical trial. The investigators aim to measure the effect of standardized acupuncture treatment, three repeated sessions, on infant colic in a randomized singe blinded prospective multi-center study, starting September 2009. The study will be done in thirteen locations in Norway by specialists in General Practice trained in acupuncture.

The investigators intend to include a total of 130 patients, 65 in the intervention group and 65 in the control group.

ELIGIBILITY:
Inclusion Criteria:

* Infants under 3 months of age with birth weight over 2500 g and/or over 36th week of gestation.
* Further fulfilling Wessel et al criteria for infant colic: "Paroxystic uncontrollable crying in an otherwise healthy child under 3 months of age, and with more than 3 hours of crying per day for more than 3 days a week for more than 3 weeks."

Exclusion Criteria:

* Infants over 3 months of age with birth weight under 2500 g and/or under 36th week of gestation.
* Not fulfilling Wessel et al criteria for infant colic: "Paroxystic uncontrollable crying in an otherwise healthy child under 3 months of age, and with more than 3 hours of crying pr.day for more than 3 days a week for more than 3 weeks."

Ages: 3 Weeks to 3 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2009-09; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Holgeir Skjeie, MD, Principal Investigator — Institute of Primary Care and Community Health, Faculty of Medicine, University of Oslo
Locations (1):
- Institute of Primary Care and Community Health, Faculty of Medicine, University of Oslo., Oslo, Norway

REFERENCES:
- [Result] Skjeie H, Skonnord T, Fetveit A, Brekke M. Acupuncture for infantile colic: a blinding-validated, randomized controlled multicentre trial in general practice. Scand J Prim Health Care. 2013 Dec;31(4):190-6. doi: 10.3109/02813432.2013.862915. Epub 2013 Nov 15. PMID 24228748
- [Derived] Skjeie H, Skonnord T, Fetveit A, Brekke M. A pilot study of ST36 acupuncture for infantile colic. Acupunct Med. 2011 Jun;29(2):103-7. doi: 10.1136/aim.2010.003590. Epub 2011 Mar 29. PMID 21450707

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The inclusion period was from September 2009 to December 2012.13 GP offices participated. The participating doctors were all GP specialists with a minimum of 300 hours of acupuncture education and fi ve years of practising acupuncture. The patients fulfi lled Wessel ' s criteria and were born at full term.
Pre-assignment Details: 113 pasients were recruited. 23 were excluded beacuse of spontanous improving of symptoms, transportation problems, change of mind regarding participation.90 patients were randomized. 79 crying diaries and 84 interviews were analysed.
Groups:
- Acupuncture: Infants born after 36th week of gestation and weighing over 2500 grams at birth, and who qualify according to Wessels definition:
  Paroxystical, uncontrolled crying in an otherwise healthy child under 3 months of age, and with more than 3 hours of crying 3 days per week for 3 weeks.
  Acupuncture with Seirin 020x15 mm sterile acupuncture needle : Bilateral insertion of a Seirin 020x15mm sterile acupuncture needle to a depth of 12mm for 30 seconds during 3 consecutive working days at the WHO designated acupuncture point St36.
Period: Overall Study
Arm/Group | Acupuncture | Control
Started | 45 | 45
Completed | 38 | 41
Not Completed | 7 | 4
Not completed — Lost to Follow-up | 6 | 3
Not completed — intercurrent febrile illness | 1 | 1

BASELINE CHARACTERISTICS:
Population: We analyzed 79 crying diaries and 84 interviews. The baseline characteristics, except crying time is based on the 84 interviews where we had complete data. The crying time is based on the 79 crying diaries
Groups:
- Acupuncture: Infants born after 36th week of gestation and weighing over 2500 grams at birth, and who qualify according to Wessels definition:
  Paroxystical, uncontrolled crying in an otherwise healthy child under 3 months of age, and with more than 3 hours of crying 3 days per week for 3 weeks.
  Acupuncture with Seirin 020x15 mm sterile acupuncture needle : Bilateral insertion of a Seirin 020x15mm sterile acupuncture needle to a depth of 12mm for 30 seconds during 3 consecutive working days at the WHO designated acupuncture point St36.
  The baseline characteristics of age and gender are based on the 84 collected interviews, while the crying time baseline units are based on the 79 collected crying time diaries. This is why numbers differ from the Participant Flow module. Only 79 participants were analyzed for crying time.
- Control: Infants born after 36th week of gestation and weighing over 2500 grams at birth, and who qualify according to Wessels definition:
  Paroxystical, uncontrolled crying in an otherwise healthy child under 3 months of age, and with more than 3 hours of crying 3 days per week for 3 weeks.
  The Control group will have no intervention.
  The baseline characteristics of age and gender are based on the 84 collected interviews, while the crying time baseline units are based on the 79 collected crying time diaries. This is why numbers differ from the Participant Flow module. Only 79 participants were analyzed for crying time.
- Total: Total of all reporting groups
Arm/Group | Acupuncture | Control | Total
Number analyzed (Participants) | 44 | 40 | 84
Age, Continuous [Mean (Full Range); unit: weeks] | 6 [3 to 13] | 6 [3 to 9] | 6 [3 to 13]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 20 | 42
  Male | 22 | 20 | 42
baseline crying time in minutes [Mean (Full Range); unit: crying time in minutes] — Daily accumulative crying time pr 24 hours as measured in a crying registration diary by the parents and returned to the investigators after the registration period.
  crying time in minutes | 220 [80 to 394] | 212 [0 to 353] | 216 [0 to 394]

OUTCOME MEASURES:

1. Primary Outcome: Change in Crying Time Per 24 Hour Period.
Description: Crying time per 24 hour period at baseline and post treatment
Time Frame: 6 time points measured: First, second and third intervention day, one day after last intervention, one week after last intervention and one month after last intervention. All time points measured in 24 hours.
Measure: Mean (95% Confidence Interval); unit: minutes crying time pr 24 hour
Arm/Group | Acupuncture | Control
Number analyzed (Participants) | 38 | 41
minutes crying time pr 24 hour
  Day 1 and 2-baseline | 220 [195 to 245] | 212 [183 to 241]
  Day 3- 1 intervention day | 230 [180 to 281] | 186 [142 to 230]
  Day 4- 2 intervention day | 180 [128 to 232] | 185 [131 to 239]
  Day 5- 3 intervention day | 129 [97 to 162] | 167 [123 to 211]
  Day 6- 1 day after intervention | 120 [94 to 145] | 142 [106 to 179]
  Day12- 1 week after intervention | 121 [79 to 164] | 120 [91 to 149]
  Day 33- 4 weeks after intervention | 89 [55 to 123] | 97 [67 to 126]

2. Secondary Outcome: Parents Evaluation of Benefit to the Child.
Description: Parents subjective assessment of the childs condition, on a 5 point scale, with 1 being worse and 5 being completely well.
  The numbers are the actual evaluations on the time specified.
Time Frame: 5 days, 1 , and 4 weeks after the first treatment
Population: The differences in numbers on parents evaluation of the childs condition (37 and 38) is due to one location assistant not reporting back on these results. Thus the number of interviews, 84, and secondary outcome data is not consistent with the numbers in the flow diagram.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Acupuncture | Control
Number analyzed (Participants) | 38 | 37
units on a scale
  Improvement day 5 | 2.87 (0.844) | 2.78 (0.917)
  Improvement day 12 | 3.62 (0.861) | 3.27 (0.902)
  Improvement day 33 | 4.03 (0.885) | 3.51 (1.146)

ADVERSE EVENTS:
Arm/Group | Acupuncture | Control
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/45
Other Adverse Events (participants affected / at risk) | 2/45 | 8/45
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Acupuncture (N=45) | Control (N=45)
Hickup (Gastrointestinal disorders) | 1 (1) | 0 (0)
Increased regurgitation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small Hematoma (General disorders) | 0 (0) | 1 (1)
Crying (General disorders) | 0 (0) | 1 (1)
Restlessness (General disorders) | 0 (0) | 1 (1)
Excessive stools (Gastrointestinal disorders) | 0 (0) | 1 (1)
Frequent defecation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Light sedation (General disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Unease (General disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Our choice of acupuncture points and technique could be inferior to other more potent acupuncture approaches.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No